CLINICAL TRIAL: NCT02498210
Title: IVM Treatment in Patients With Low Ovarian Response. Does it Improve IVF Outcome or May it Cause Activation of Ovarian Follicles and Increase the Chances of Success in the Following IVF Cycle?
Brief Title: IVM for Patients With Low Ovarian Response. Does it Improve IVFoutcomes and Does it Improve the Following IVF Cycle?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1604-EM-CTIL
Record Dates: First submitted 2015-05-31; First posted 2015-07-15 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Infertility Female
Keywords: IVM; HIPPO signaling
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVF after IVM (Experimental): If the patients will not concive during the IVM cycle . results of this following IVF cycle will be compared to the initial IVF preformance
  Intervention : In Vitro Maturation Procedure
  Interventions: Other: In Vitro Maturation Procedure

INTERVENTIONS:
Other: In Vitro Maturation Procedure — POR patients will be treated in IVM cycle. After baseline evaluation on day 3, 150 IU/day recombinant FSH or HMG will be added for 3 days. A second evaluation will be performed on day 6 of the menstrual cycle. An injection of 10,000 IU hCG (Pregnyl; Organon, Oss, Holland) or Ovitrelle 250mcg (Merck Serono ) will be administered subcutaneously when the endometrial thickness will be ≥6 mm and the leading follicle will be at least 12 mm. Oocyte retrieval will be performed under ultrasound guidance with a 19G single-lumen aspiration needle (Cook; Queensland, Australia). The follicular fluid will be collected in culture tubes containing follicle flush buffer (Cook) with 2 IU/ml heparin. All aspirates were filtered to identify additional oocytes

SUMMARY:
Poor ovarian response (POR) is one of the major therapeutic challenges in in vitro fertilization. Several therapeutic approaches for POR have been explored; yet, a single effective strategy has not yet been established. Recently, a live birth was reported after ovarian cortex fragmentation and in vitro disruption of the Hippo signaling pathway and activation of Akt signaling. During IVM procedure increased mechanical stimulation of the ovarian cortex takes place. , with the consequent disruption of the Hippo signaling pathway. Our aim is to investigate whether the mechanical manipulation and triggering of ovarian cortex caused by IVM can cause ovarian follicular activation and recruitment by the mechanisms mentioned above. Thus stimulation in the following regular IVF cycle will result in improved ovarian response and increased oocytes yield

DETAILED DESCRIPTION:
IVM treatment in patients with low ovarian response. Does it improve IVF outcome or may it cause activation of ovarian follicles and increase the chances of success in the following IVF cycle?

Scientific background:

Poor ovarian response (POR) is one of the major therapeutic challenges in in vitro fertilization. The prevalence of poor responders patients varies in the literature between 9 and 24%, however due to the increase in childbearing age it is expected to be one of the main infertility cause. Failure to respond adequately to standard protocols and to recruit adequate follicles results in decreased oocyte production, cycle cancellation and, overall, it is associated with a significantly diminished probability of pregnancy Several therapeutic approaches for POR have been explored; yet, a single effective strategy has not yet been established. Previously it was shown that mechanical manipulation on ovarian cortex such as ovarian wedge resection or ovarian "drilling" by diathermy or laser, induced follicle growth in polycystic ovarian syndrome (PCOS) patient.

Recently, a live birth was reported after ovarian cortex fragmentation and in vitro disruption of the Hippo signaling pathway and activation of Akt signaling. The treated ovarian fragments were grafted back to the patient and after follicle growth, retrieval of mature eggs, in vitro fertilization and embryo transfer; a healthy baby was delivered. The Hippo signaling pathway is essential to maintain optimal organ size and is conserved in all metazoan animals [6-8]. In this study it was shown that ovarian fragmentation increased actin polymerization and disrupted Hippo signaling by decreasing phosphorylated Yes-associated protein (pYAP) levels together with increased nuclear localization of YAP, leading to increased expression of CCN growth factors genes and BIRC apoptosis inhibitors. Secreted CCN2 and related factors promoted follicle growth

Genes involved in ovarian fragmentation, Hippo signaling, and follicle growth is important for ovarian physiology and pathophysiology. Ovarian fragmentation led to changes in intercellular tension and facilitated the conversion of G-actin to F-actin. Subsequent disruption of Hippo signaling decreased pYAP to total YAP ratios, leading to increased expression of downstream CCN growth factors and BIRC apoptosis inhibitors

In vitro maturation (IVM) has been practiced in a clinical setting for over a decade. It has been suggested as an alternative to conventional IVF for minimizing the risk of the ovarian hyperstimulation syndrome (OHSS) in patients with the PCOS. Recently, IVM has been proposed as the method for patients undergoing anticancer treatment, particularly for women who require rapid fertility preservation [9] or face the risk of estrogen-sensitive cancer recurrence involve. Although IVM has been applied to IVF poor responders with equivocal results, several researchers have shown benefits in IVM in women who have low ovarian response.

For the purpose of IVM, oocytes are retrieved from ovarian follicles as small as 4-5mm in diameter, under ultrasound guidance with a single-lumen thinner aspiration needle. The aspiration pressure is reduced compared to regular IVF. Therefore, multiple needle punctures are needed because lower aspiration pressures are used and bloody aspirates may block the thin needle lumen. Because immature oocytes are enclosed in tightly packed cumulus cells, curettage of the follicle wall is needed to dislodge the cumulus oocyte complex. All leads to the fact that during IVM procedure increased mechanical stimulation of the ovarian cortex takes place, with the consequent disruption of the Hippo signaling pathway.

Hypothesis and aims Our aim is to investigate whether the mechanical manipulation and triggering of ovarian cortex caused by IVM can cause ovarian follicular activation and recruitment by the mechanisms mentioned above. Thus stimulation in the following regular IVF cycle will result in improved ovarian response and increased oocytes yield.

Materials and Methods Patients Prospective cohort study on POR patients. Twenty five POR patients will be selected based on the bologna criteria and all patients will have at least one documented POR cycle.

IVM protocol POR patients will be treated in IVM cycle according to our IVF unit protocol, using FSH-priming . Briefly, a baseline evaluation that included a hormonal profile and an ultrasound scan was performed on day 3 of the menstrual cycle. On day 3, 150 IU/day recombinant FSH was added for 3 days. A second evaluation was performed on day 6 of the menstrual cycle. An injection of 10,000 IU hCG (Pregnyl; Organon, Oss, Holland) was administered subcutaneously when the endometrial thickness will be ≥6 mm and the leading follicle will be at least 12 mm. Oocyte retrieval will be performed under ultrasound guidance with a 19G single-lumen aspiration needle (Cook; Queensland, Australia) with a reduced aspiration pressure of 7.5 kPa. The follicular fluid will be collected in culture tubes containing follicle flush buffer (Cook) with 2 IU/ml heparin. Because of the difficulty in identifying compacted oocyte complexes, all aspirates were filtered to identify the additional oocytes.

In-Vitro Oocyte Maturation Germinal vesicles and M1 oocytes will be cultured in IVM medium (Sage; CT, USA) supplemented with 75 IU FSH and 75IU luteinizing hormone (LH; Ferring, Keil, Germany) and checked for maturity between 24-48 hours after culture. Mature oocytes were will be denuded of the granulosa cells and fertilized by intracytoplasmic sperm injection (ICSI). After ICSI, the oocytes will be transferred into IVF medium. Fertilization will be assessed 18 hours after ICSI by examining the oocytes for the appearance of two distinct pronuclei (2PN) and the extrusion of two polar bodies.

IVF protocol Following the IVM treatment, if the patient failed to conceive, she will be offered a conventional IVF treatment, using the same controlled ovarian hyperstimulation protocol, as in her previous IVF treatment (prior to the IVM cycle). Each patient will serve as her own control.

Outcome measurements Outcome measurements will include controlled ovarian hyperstimulation variables, number of retrieved oocytes, mature oocytes on the day of the aspiration, fertilization rate, embryos quality and number of embryos transferred.

ELIGIBILITY:
Inclusion Criteria:

Poor ovarian response IVF cycle

Exclusion Criteria:

Normal ovarian response

-

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes | 3 month
  IVF cycle after IVM results will be compared to the IVF cycle with poor ovarian response

CONTACTS AND LOCATIONS:
Overall Officials: Ettie Maman, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Kiryat Ono, Israel

REFERENCES:
- [Background] Venetis CA, Kolibianakis EM, Tarlatzi TB, Tarlatzis BC. Evidence-based management of poor ovarian response. Ann N Y Acad Sci. 2010 Sep;1205:199-206. doi: 10.1111/j.1749-6632.2010.05665.x. PMID 20840273
- [Background] Shanbhag S, Aucott L, Bhattacharya S, Hamilton MA, McTavish AR. Interventions for 'poor responders' to controlled ovarian hyperstimulation (COH) in in-vitro fertilisation (IVF). Cochrane Database Syst Rev. 2007 Jan 24;(1):CD004379. doi: 10.1002/14651858.CD004379.pub2. PMID 17253503
- [Background] STEIN IF Sr. The management of bilateral polycystic ovaries. Fertil Steril. 1955 May-Jun;6(3):189-205. doi: 10.1016/s0015-0282(16)31980-x. No abstract available. PMID 14380378
- [Background] Farquhar C, Brown J, Marjoribanks J. Laparoscopic drilling by diathermy or laser for ovulation induction in anovulatory polycystic ovary syndrome. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD001122. doi: 10.1002/14651858.CD001122.pub4. PMID 22696324
- [Background] Kawamura K, Cheng Y, Suzuki N, Deguchi M, Sato Y, Takae S, Ho CH, Kawamura N, Tamura M, Hashimoto S, Sugishita Y, Morimoto Y, Hosoi Y, Yoshioka N, Ishizuka B, Hsueh AJ. Hippo signaling disruption and Akt stimulation of ovarian follicles for infertility treatment. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17474-9. doi: 10.1073/pnas.1312830110. Epub 2013 Sep 30. PMID 24082083
- [Background] Dong J, Feldmann G, Huang J, Wu S, Zhang N, Comerford SA, Gayyed MF, Anders RA, Maitra A, Pan D. Elucidation of a universal size-control mechanism in Drosophila and mammals. Cell. 2007 Sep 21;130(6):1120-33. doi: 10.1016/j.cell.2007.07.019. PMID 17889654
- [Background] Hergovich A. Mammalian Hippo signalling: a kinase network regulated by protein-protein interactions. Biochem Soc Trans. 2012 Feb;40(1):124-8. doi: 10.1042/BST20110619. PMID 22260677
- [Background] Maman E, Meirow D, Brengauz M, Raanani H, Dor J, Hourvitz A. Luteal phase oocyte retrieval and in vitro maturation is an optional procedure for urgent fertility preservation. Fertil Steril. 2011 Jan;95(1):64-7. doi: 10.1016/j.fertnstert.2010.06.064. Epub 2010 Aug 5. PMID 20688325
- [Background] Li J, Xu Y, Zhou G, Guo J, Xin N. Natural cycle IVF/IVM may be more desirable for poor responder patients after failure of stimulated cycles. J Assist Reprod Genet. 2011 Sep;28(9):791-5. doi: 10.1007/s10815-011-9597-6. Epub 2011 Jun 22. PMID 21695516
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041